CLINICAL TRIAL: NCT03019146
Title: Exploring Time-efficient Strategies to Improve Fitness for Surgery in Older Adults
Acronym: eHHH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Nottingham (Other)
Collaborators: The Royal College of Surgeons of England (Other); The Dunhill Medical Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A12092016
Record Dates: First submitted 2017-01-04; First posted 2017-01-12 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Perioperative Hypertension; Hypertension
Keywords: Prehabilitation
MeSH Terms: conditions — Hypertension | interventions — High-Intensity Interval Training; Exercise; Ischemic Preconditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- High Intensity Interval Training (HIIT) (Experimental): 3 x 15 minute sessions per week for 6 weeks. Sessions include 5x intervals of cycling at 110% of Wmax derived from CPET, interspersed with 90s rest periods of unloaded cycling.
  Interventions: Other: HIIT
- Isometric Handgrip (HOLD) (Experimental): 3x 15 minute sessions per week for 6 weeks Sessions include 4x intervals of 2minutes isometric handgrip contraction of dominant arm at 30% Maximal voluntary contraction, interspersed with 2minute rest periods
  Interventions: Other: HOLD
- Remote Ischaemic Preconditioning (HUG) (Experimental): 3x 15 minute sessions per week for 6 weeks. Sessions include 3x intervals of 3 minutes of arm ischaemia (blood pressure cuff inflated to 200mmHg on dominant arm) interspersed with 3 minute rest periods.
  Interventions: Other: HUG
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: HIIT
  Other Names: High intensity Interval training
  Arms: High Intensity Interval Training (HIIT)
Other: HOLD
  Other Names: Isometric exercise; Isometric handgrip
  Arms: Isometric Handgrip (HOLD)
Other: HUG
  Other Names: Remote ischaemic preconditioning; Ischaemic preconditioning
  Arms: Remote Ischaemic Preconditioning (HUG)

SUMMARY:
The incidence of conditions requiring surgical intervention increases with age, however there is a reported decline in the rates of elective surgical procedures in those over 65. This is associated with older patients being described as "less fit" and more at risk of postoperative complications, leading to decreased provision of surgical care to those at need. Exercise interventions have the potential to reverse some of the decline in cardiovascular fitness associated with aging and improve the elderly's' "fitness for surgery" and potentially allow increased access to surgical care for those most in need of it.

DETAILED DESCRIPTION:
The percentage of people aged >65 y in the United Kingdom increased from 15% in 1985 to 17% in 2010, an increase of 1.7 million people. One age-associated physiological change is the reduction in vascular function that is observed, both at the levels of the large arteries and the muscle microvasculature. In itself this vascular dysfunction is associated with reduced aerobic performance. Cardiorespiratory fitness (marked by aerobic performance) has been shown to be an independent predictor of postoperative mortality, which provides more accurate prognostic information than age alone. In contrast, physical activity can reverse elements of pathophysiology associated with these conditions, including vascular dysfunction. Nonetheless, major roadblocks to exercise as a strategy to combat age-associated vascular dysfunction and associated conditions exist, namely: i) poor exercise tolerance, ii) "lack of time", iii) age-related mobility impairments, and iv) exercise resistance.

The aim of this study is to investigate whether if novel low-volume, time-efficient training strategies can improve indices of vascular health and cardiorespiratory performance in older individuals with a view towards improving their fitness for surgery. Numerous studies have demonstrated that periods of supervised exercise training effectively improve indices of cardiorespiratory (blood pressure, aerobic capacity and blood lipids and vascular function. However, the majority of these studies were conducted using high-volume continuous submaximal aerobic training (e.g. 50-65% VO2max for 30-60 min) or moderate to high volume progressive weight training. This research group have recently shown the efficacy of a time-efficient exercise strategy known as HIIT - High Intensity Interval Training, for improving VO2 max and muscle mass in young individuals with heightened metabolic disease risk and also demonstrated significant improvements in VO2 max comparable to classic aerobic exercise training using several different time-efficient HIIT protocols. However, despite the potential benefits of HIIT, not least its 70-80% reduction in required time-commitment compared to current WHO guidelines, it does have limitations, particularly for an older population where physical (mobility/joint) and/or socio-economic (transport/gym access/equipment purchase) barriers may render it ineffective and/or unachievable.

Alternative interventions for prevention or treatment of age-associated vascular dysfunction could be provided by isometric handgrip training (IHG) or remote ischaemic pre-conditioning (RIPC), both of which have a similar low time-commitment compared to HIIT but are less strenuous, have potential as home-based interventions, and require only inexpensive equipment. IHG has been demonstrated to improve resting blood pressure in both normotensive and medicated hypertensive populations to a similar or greater extent as classic aerobic exercise training. However, the effects of IHG on other vascular (e.g. limb, brain and muscle microvascular blood flow) or cardio-respiratory parameters (VO2 max, heart rate (resting/recovery), exercise tolerance) have not been assessed. Similarly, although RIPC has recently been shown to improve maximal athletic cardio-respiratory performance and vascular function in young subjects, no work to date has explored the efficacy of chronic RIPC on indices of health or vascular function in older individuals.

Therefore, the aims of this project are to:

(i) Assess the efficacy of 6 weeks HIT, IHG and RIPC for improving indices of cardio-respiratory, vascular and metabolic function in older subjects as a means of improving fitness for surgery.

(ii) Explore the concept of "exercise resistance" in relation to HIT, IHG and RIPC by:

1. Assessing if the same degree of response heterogeneity exists for the three time-efficient training modes employed in this study as has been reported for classic resistance and aerobic exercise training
2. Assessing if a "non-responder" for one index (i.e., resting blood pressure or leg blood flow) is a non-responder for all other indices

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer aged 65-85

Exclusion Criteria:

* • Current participation in a formal exercise regime

  * A BMI < 18 or > 32 kg·m2
  * Active cardiovascular disease:

    * uncontrolled hypertension (BP > 160/100),
    * angina,
    * heart failure (class III/IV),
    * Significant arrhythmia,
    * right to left cardiac shunt,
    * recent cardiac event
  * Taking beta-adrenergic blocking agents,
  * Cerebrovascular disease:

    * previous stroke,
    * aneurysm (large vessel or intracranial)
    * epilepsy
  * Respiratory disease including:

    * pulmonary hypertension,
    * Significant COPD,
    * Uncontrolled asthma,
  * Metabolic disease:

    * hyper and hypo parathyroidism,
    * untreated hyper and hypothyroidism,
    * Cushing's disease,
    * type 1 or 2 diabetes
  * Active inflammatory bowel or renal disease
  * Malignancy
  * Clotting dysfunction
  * Significant Musculoskeletal or neurological disorders
  * Family history of early (<55y) death from cardiovascular disease
  * Known sensitivity to Sonovue

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in resting systolic blood pressure | 6 weeks
  Measured in seated position using oscillometry, mean value of 3 recordings, measured according to British Society of Hypertension Guidelines 2013.

SECONDARY OUTCOMES:
Change in resting diastolic blood pressure | 6 weeks
  Measured using a ramp incremental exercise test on a cycle ergometer.
Ambulatory blood pressure | 6 weeks
  Ambulatory blood pressure
V02 Peak | 6 weeks
  Measured using a ramp incremental exercise test on a cycle ergometer.
Anaerobic threshold | 6 weeks
  Measured using a ramp incremental exercise test on a cycle ergometer.
Body fat percentage | 6 weeks
  Measured by dual energy X-ray absorptiometry
Total body lean mass | 6 weeks
  Measured by dual energy X-ray absorptiometry
Change in common femoral artery blood flow | 6 weeks
  Measured by duplex ultrasound on non-dominant leg in response to 6 unilateral leg extensions at 50% 1 repetition maximum
Change in Vastus lateralis microvascular blood flow | 6 weeks
  Measured by contrast enhanced ultrasound on the dominant leg in response to 6 unilateral leg extensions at 50% 1 repetition maximum
Flow-mediated dilatation | 6 weeks
Heart rate recovery post exercise | 6 weeks
  Change in heart rate after exercise from peak over time
Blood pressure recovery post exercise | 6 weeks
  Change in blood pressure after exercise from peak over time
Area under concentration curve for serum Glucose | 6 weeks
  Measured from a 3 hour oral glucose tolerance test
Area under concentration curve for serum Insulin | 6 weeks
  Measured from a 3 hour oral glucose tolerance test
Matsuda Index of insulin sensitivity | 6 weeks
  Measured from a 3 hour oral glucose tolerance test
Cederholm Index of insulin sensitivity | 6 weeks
  Measured from a 3 hour oral glucose tolerance test
Homeostatic Model Assessment of Insulin Resistance | 6 weeks
  Measured from fasting plasma samples, taken before a 3 hour oral glucose tolerance test
Fasting Serum Cholesterol | 6 weeks
Fasting serum triglyceride | 6 weeks
Time to failure, cycling at 50% maximum power achieved during CPET | 6 weeks
Handgrip maximum voluntary contraction | 6 weeks
  Measured using a handgrip dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- University Of Nottingham, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] LaRocca TJ, Hearon CM Jr, Henson GD, Seals DR. Mitochondrial quality control and age-associated arterial stiffening. Exp Gerontol. 2014 Oct;58:78-82. doi: 10.1016/j.exger.2014.07.008. Epub 2014 Jul 14. PMID 25034910
- [Background] Phillips BE, Atherton PJ, Varadhan K, Limb MC, Wilkinson DJ, Sjoberg KA, Smith K, Williams JP. The effects of resistance exercise training on macro- and micro-circulatory responses to feeding and skeletal muscle protein anabolism in older men. J Physiol. 2015 Jun 15;593(12):2721-34. doi: 10.1113/JP270343. Epub 2015 May 14. PMID 25867865
- [Background] Gonzalez-Alonso J, Calbet JA. Reductions in systemic and skeletal muscle blood flow and oxygen delivery limit maximal aerobic capacity in humans. Circulation. 2003 Feb 18;107(6):824-30. doi: 10.1161/01.cir.0000049746.29175.3f. PMID 12591751
- [Background] Snowden CP, Prentis J, Jacques B, Anderson H, Manas D, Jones D, Trenell M. Cardiorespiratory fitness predicts mortality and hospital length of stay after major elective surgery in older people. Ann Surg. 2013 Jun;257(6):999-1004. doi: 10.1097/SLA.0b013e31828dbac2. PMID 23665968
- [Background] Iwasaki K, Zhang R, Zuckerman JH, Levine BD. Dose-response relationship of the cardiovascular adaptation to endurance training in healthy adults: how much training for what benefit? J Appl Physiol (1985). 2003 Oct;95(4):1575-83. doi: 10.1152/japplphysiol.00482.2003. Epub 2003 Jun 27. PMID 12832429
- [Background] Wilmore JH, Green JS, Stanforth PR, Gagnon J, Rankinen T, Leon AS, Rao DC, Skinner JS, Bouchard C. Relationship of changes in maximal and submaximal aerobic fitness to changes in cardiovascular disease and non-insulin-dependent diabetes mellitus risk factors with endurance training: the HERITAGE Family Study. Metabolism. 2001 Nov;50(11):1255-63. doi: 10.1053/meta.2001.27214. PMID 11699041
- [Background] Vollaard NB, Constantin-Teodosiu D, Fredriksson K, Rooyackers O, Jansson E, Greenhaff PL, Timmons JA, Sundberg CJ. Systematic analysis of adaptations in aerobic capacity and submaximal energy metabolism provides a unique insight into determinants of human aerobic performance. J Appl Physiol (1985). 2009 May;106(5):1479-86. doi: 10.1152/japplphysiol.91453.2008. Epub 2009 Feb 5. PMID 19196912
- [Background] Kraus WE, Houmard JA, Duscha BD, Knetzger KJ, Wharton MB, McCartney JS, Bales CW, Henes S, Samsa GP, Otvos JD, Kulkarni KR, Slentz CA. Effects of the amount and intensity of exercise on plasma lipoproteins. N Engl J Med. 2002 Nov 7;347(19):1483-92. doi: 10.1056/NEJMoa020194. PMID 12421890
- [Background] Santos-Parker JR, LaRocca TJ, Seals DR. Aerobic exercise and other healthy lifestyle factors that influence vascular aging. Adv Physiol Educ. 2014 Dec;38(4):296-307. doi: 10.1152/advan.00088.2014. PMID 25434012
- [Background] Seals DR. Edward F. Adolph Distinguished Lecture: The remarkable anti-aging effects of aerobic exercise on systemic arteries. J Appl Physiol (1985). 2014 Sep 1;117(5):425-39. doi: 10.1152/japplphysiol.00362.2014. Epub 2014 May 22. PMID 24855137
- [Background] Kraus WE, Torgan CE, Duscha BD, Norris J, Brown SA, Cobb FR, Bales CW, Annex BH, Samsa GP, Houmard JA, Slentz CA. Studies of a targeted risk reduction intervention through defined exercise (STRRIDE). Med Sci Sports Exerc. 2001 Oct;33(10):1774-84. doi: 10.1097/00005768-200110000-00025. PMID 11581566
- [Background] Church TS, Earnest CP, Skinner JS, Blair SN. Effects of different doses of physical activity on cardiorespiratory fitness among sedentary, overweight or obese postmenopausal women with elevated blood pressure: a randomized controlled trial. JAMA. 2007 May 16;297(19):2081-91. doi: 10.1001/jama.297.19.2081. PMID 17507344
- [Background] Phillips B, Williams J, Atherton P, Smith K, Hildebrandt W, Rankin D, Greenhaff P, Macdonald I, Rennie MJ. Resistance exercise training improves age-related declines in leg vascular conductance and rejuvenates acute leg blood flow responses to feeding and exercise. J Appl Physiol (1985). 2012 Feb;112(3):347-53. doi: 10.1152/japplphysiol.01031.2011. Epub 2011 Oct 13. PMID 21998269
- [Background] Metcalfe RS, Babraj JA, Fawkner SG, Vollaard NB. Towards the minimal amount of exercise for improving metabolic health: beneficial effects of reduced-exertion high-intensity interval training. Eur J Appl Physiol. 2012 Jul;112(7):2767-75. doi: 10.1007/s00421-011-2254-z. Epub 2011 Nov 29. PMID 22124524
- [Background] Garg R, Malhotra V, Kumar A, Dhar U, Tripathi Y. Effect of isometric handgrip exercise training on resting blood pressure in normal healthy adults. J Clin Diagn Res. 2014 Sep;8(9):BC08-10. doi: 10.7860/JCDR/2014/8908.4850. Epub 2014 Sep 20. PMID 25386422
- [Background] Millar PJ, McGowan CL, Cornelissen VA, Araujo CG, Swaine IL. Evidence for the role of isometric exercise training in reducing blood pressure: potential mechanisms and future directions. Sports Med. 2014 Mar;44(3):345-56. doi: 10.1007/s40279-013-0118-x. PMID 24174307
- [Background] Jean-St-Michel E, Manlhiot C, Li J, Tropak M, Michelsen MM, Schmidt MR, McCrindle BW, Wells GD, Redington AN. Remote preconditioning improves maximal performance in highly trained athletes. Med Sci Sports Exerc. 2011 Jul;43(7):1280-6. doi: 10.1249/MSS.0b013e318206845d. PMID 21131871
- [Background] Jones H, Hopkins N, Bailey TG, Green DJ, Cable NT, Thijssen DH. Seven-day remote ischemic preconditioning improves local and systemic endothelial function and microcirculation in healthy humans. Am J Hypertens. 2014 Jul;27(7):918-25. doi: 10.1093/ajh/hpu004. Epub 2014 Mar 13. PMID 24627443
- See also: Office for National Statistics; Population Ageing in the United Kingdom, its Constituent Countries and the European Union — http://webarchive.nationalarchives.gov.uk/20160105160709/http://www.ons.gov.uk/ons/dcp171776_258607.pdf